CLINICAL TRIAL: NCT00573209
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation Treatment for Erectile Dysfunction.
Brief Title: Energy Specific Far Infrared Radiation Treatment for Erectile Dysfunction
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder & President, GAAD Medical Research Institute inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-EDS-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Erectile Dysfunction
Keywords: Impotence; Male Impotence; Male Sexual Impotence
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Radiation: Far Infrared Radiation

INTERVENTIONS:
Radiation: Far Infrared Radiation — Far Infrared Radiation (5μm to 20μm wavelength) for 30 to 40 minutes each session.

SUMMARY:
A preliminary study to determine the possibility of using far infrared (FIR) radiation to treat impotency.

DETAILED DESCRIPTION:
Erectile dysfunction is characterized by the regular or repeated inability to obtain or maintain an erection. Erection depends on a complex interaction of psychological, neural, vascular and endocrine factors.

We are proposing a non-drug and a non-invasive radiation treatment for the enhancement of erection.

ELIGIBILITY:
Inclusion Criteria:

* Persons with erection challenges

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation on erectile dysfunction. | 1 year

SECONDARY OUTCOMES:
The effect of far infrared radiation on other male conditions like prostate cancer | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Study Director — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Chair — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Mississauga, Ontario, Canada